CLINICAL TRIAL: NCT04149210
Title: FLuorometholone as Adjunctive MEdical Therapy for TT Surgery (FLAME) Trial
Acronym: FLAME
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Collaborators: University of Pennsylvania (Other); London School of Hygiene and Tropical Medicine (Other); Berhan Public Health and Eye Care Consultancy PLC (Other); The Fred Hollows Foundation, Ethiopia (Unknown); The Fred Hollows Foundation, Australia (Unknown)
Responsible Party: Principal Investigator, John Harold Kempen, Professor, Director of Epidemiology for Ophthalmology, Massachusetts Eye and Ear Infirmary
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019P002286
Record Dates: First submitted 2019-10-12; First posted 2019-11-04 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Trachomatous Trichiasis (TT); Eye Diseases; Eyelid Diseases; Trachomatous; Trichiasis
Keywords: fluorometholone 0.1%; trachomatous trichiasis; Eye Diseases; Eyelid Diseases; trachomatous; trichiasis; FLAME; TT Surgery
MeSH Terms: conditions — Eye Diseases; Eyelid Diseases; Trichiasis | interventions — Fluorometholone; Lubricant Eye Drops

STUDY DESIGN:
Intervention Model Description: This is a 1:1 randomized, double-masked, placebo controlled clinical trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patients, surgeons, and study staff at field site are masked to the assigned treatment group of the subject.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fluorometholone (Experimental): Fluorometholone 0.1% eyedrops, one drop twice daily for four weeks
  Interventions: Drug: Fluorometholone 0.1% Oph Susp
- Artificial Tears (Placebo Comparator): one drop two times daily for four weeks
  Interventions: Drug: Artificial Tears

INTERVENTIONS:
Drug: Fluorometholone 0.1% Oph Susp — fluorometholone 0.1% one drop twice daily for four weeks, beginning with one drop just before trachomatous trichiasis surgery on the upper lid.
  Other Names: FML
  Arms: fluorometholone
Drug: Artificial Tears — Artificial tears (placebo) given one drop twice daily for four weeks, beginning with one drop just prior to trachomatous trichiasis surgery on the upper lid.
  Other Names: Placebo
  Arms: Artificial Tears

SUMMARY:
This study aims :

* To assess the efficacy of fluorometholone 0.1% one drop twice daily for four weeks in reducing the incidence of post-operative trachomatous trichiasis (TT) when given as adjunctive therapy with TT surgery in the programmatic setting
* To assess whether such treatment is sufficiently safe for wide-scale implementation in TT programs.
* To estimate the costs of adding fluorometholone 0.1% treatment to TT surgery per case of postoperative TT averted, and to characterize the value of such treatment under a range of plausible health economic circumstances

DETAILED DESCRIPTION:
The investigators are pursuing an agenda to evaluate a new potentially cost-effective approach to improving trichiasis surgery outcomes: perioperative topical anti-inflammatory therapy. Inflammation-whether induced by the trachoma disease process or surgery itself-most likely contributes to progressive cicatrization leading to failure of lid rotation surgery in a clinically important proportion of TT cases. The investigators hypothesize that adjunctive topical fluorometholone therapy following trichiasis surgery will reduce the risk of recurrent trichiasis and will be acceptably safe. The rationale for the efficacy aspect of this hypothesis is that interruption of inflammation postoperatively would reduce postoperative scarring/contracture driven by ongoing disease-driven inflammation and/or surgically-induced inflammation thus reducing the incidence of TT recurrence (post-operative TT) and other inflammation-related outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Age 15 years or more, corresponding to the age of patients treated in the Fred Hollows Foundation/Federal Ministry of Health Program at field sites without general anesthesia.
2. One or both eyes with upper lid trachomatous trichiasis-with one or more eyelashes touching the eye or evidence of epilation, with a plan to undergo TT surgery on at least one upper eyelid.
3. Collection of all baseline data prior to randomization
4. Signed, informed consent (and assent, when applicable)

Exclusion Criteria:

1. Contraindication(s) to the use of the test articles, including a known allergy or sensitivity to the study medication (fluorometholone) or its components, and contraindication(s) to use of azithromycin
2. IOP≥22 mmHg and/or currently taking more than two ocular anti-hypertensive medications in the study eye (prior IOP-lowering surgery is acceptable; combinations of two IOP-lowering agents such as Dorzamol are considered two medications)
3. A known severe / serious ocular pathology or medical condition which may preclude study completion or increase the risk of harm in the study (e.g., suspicion of non-trachomatous active ocular infection or suspicion of glaucoma of a degree to which where an intraocular pressure spike would be vision-threatening).
4. Any condition known to be present at baseline for which it is anticipated ocular or systemic corticosteroid therapy will be required.
5. Any significant illness or condition (e.g., hypertension with systolic blood pressure≥170 mmHg and/or diastolic blood pressure≥110 mmHg) that could, in the study team's opinion, be expected to interfere with the study parameters or study conduct; or put the subject at significant risk.
6. Previous upper lid TT surgery on all eyes with upper lid TT. (If one eye has previously undergone upper lid TT surgery but another eye with upper lid TT has not, the patient may be enrolled, and only the latter eye will be counted for the primary analyses).

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2410 (Actual)
Dates: Start 2021-08-19 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative TT by one year, as determined by trained study team members | 12 months
  The primary outcome measure is the postoperative recurrence of trachomatous trichiasis (TT), defined as one or more eyelashes in the upper eyelid touching the globe or evidence of epilation (lash stubs) in the upper eyelid on examination, or a history of repeat trichiasis surgery at any time in the upper eyelid during the one year follow-up period after the baseline surgery.

SECONDARY OUTCOMES:
Efficacy Measure 1 - Entropion | 1 year
  Presence and extent of entropion of the upper eyelid
Efficacy Measure 2 - Reoperation | 1 year
  Number of study eyes undergoing reoperation for postoperative trichiasis
Efficacy Measure 3 - Lashes | 1 year
  Number and location of trichiatic lashes from the upper eyelid touching the globe
Efficacy Measure 4 - Health economic analysis | 1 year
  Marginal cost per case of postoperative trichiasis avoided (Cost-effectiveness in the use of Fluorometholone 0.1%)
Safety/adverse outcomes 1 - Corneal Opacity | 1 year
  Presence and grade of corneal opacity in study eyes
Safety/adverse outcomes 2 - Overcorrection | 1 year
  Presence of overcorrection in study eyes
Safety/adverse outcomes 3 - Eyelid Abnormalities | 1 year
  Presence of eyelid notching/eyelid contour abnormalities in study eyes
Safety/adverse outcome 4 - Lid Closure Defect | 1 year
  Presence of lid closure defect in study eyes
Safety/adverse outcomes 5 - Granuloma | 1 year
  Presence of granuloma in study eyes
Safety/adverse outcomes 6 - Pain level | 1 year
  Pain level in study eyes at one year scored from 1 (none) to 5 (extreme)
Safety/adverse outcomes 7 - IOP in mmHg | 4 weeks
  Intraocular pressure (IOP) elevation in study eyes
Safety/adverse outcomes 8 - Cataract Surgery | 1 year
  Occurrence of cataract surgery in study eyes
Safety/adverse outcomes 9 - TT in non-study eye | 1 year
  Cumulative incidence of TT in the fellow eye by one year
Safety/adverse outcomes 10 - Adverse Events | 1 year
  Adverse events attributed to study treatment
Patient-reported outcomes 1 - Patient satisfaction | 1 year
  Patient satisfaction level in regards to the trichiasis surgery outcome measured on a likert scale for satisfaction (from very dissatisfied to very satisfied)
Patient-reported outcomes 2 - Cosmetic outcome | 1 year
  Patient satisfaction level in regards to the cosmetic outcome of the trichiasis surgery measured on a likert scale for satisfaction (from very dissatisfied to very satisfied)
Patient-reported outcomes 3 - Health utility | 1 year
  Quality of life assessed using the tool EuroQol 5 Dimensions (EQ-5D) comprising mobility, self-care, usual activities, pain/discomfort and anxiety/depression dimensions and assessed on five levels from no problems to extreme problems
Additional variables 1 - Visual Acuity | 1 year
  Visual acuity with presenting correction in study eyes

CONTACTS AND LOCATIONS:
Overall Officials: John H Kempen, MD MPH MHS PhD, Study Chair — Massachusetts Eye and Ear Infirmary/Harvard Medical School
Locations (1):
- Oromia Health Bureau, Addis Ababa, Ethiopia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kempen JH, Abashawl A, Mohammed AA, Dodson S, Alemayehu W, Jin F, Gemechu A, Mengesha AA, Kumsa DA, Chen Y, McWilliams K, Tulu B, Abdela G, Megersa A, Cheru T, Mohammad G, Succar T, Bunya VY, Frick KD, Maguire MG, Burton MJ, Ying GS; FLAME Trial Research Group. Evaluation of fluorometholone as adjunctive medical therapy for trachomatous trichiasis surgery (FLAME): a parallel, double-blind, randomised controlled field trial in the Jimma Zone, Ethiopia. Lancet Glob Health. 2026 Jan 12:S2214-109X(25)00493-0. doi: 10.1016/S2214-109X(25)00493-0. Online ahead of print. PMID 41539314
- [Derived] Kempen JH, Chen Y, Abashawl A, Mohammed AA, Dodson S, Alemayehu W, Gemechu A, Mengesha AA, Kumsa DA, Succar T, McWilliams K, Jin F, Bunya VY, Maguire MG, Burton MJ, Ying GS; FLuorometholone as Adjunctive MEdical Therapy for Trachomatous Trichiasis Surgery (FLAME) Trial Research Group. Outcomes of posterior lamellar tarsal rotation vs bilamellar tarsal rotation for trachomatous trichiasis. PLoS Negl Trop Dis. 2025 Jul 30;19(7):e0013152. doi: 10.1371/journal.pntd.0013152. eCollection 2025 Jul. PMID 40737343
- [Derived] Mohammed AA, Abashawl A, Dodson S, Alemayehu W, Gemechu A, Abateneh A, Kumsa D, Succar T, Chen Y, McWilliams K, Bunya VY, Maguire MG, Burton MJ, Ying GS, Kempen JH; FLuorometholone as Adjunctive MEdical Therapy for Trachomatous Trichiasis Surgery (FLAME) Trial Research Group. The FLuorometholone as Adjunctive MEdical Therapy for Trachomatous Trichiasis Surgery (FLAME) Trial: Study Design. Ophthalmic Epidemiol. 2024 Dec;31(6):611-619. doi: 10.1080/09286586.2024.2415052. Epub 2024 Dec 10. PMID 39656933
- [Derived] Mohammed AA, Abashawl A, Dodson S, Alemayehu W, Gemechu A, Mengesha AA, Kumsa D, Succar T, Chen Y, McWilliams K, Bunya VY, Maguire MG, Burton MJ, Ying GS, Kempen JH; FLuorometholone as Adjunctive MEdical Therapy for Trachomatous Trichiasis Surgery (FLAME) Trial Research Group. The FLuorometholone as Adjunctive MEdical Therapy for Trachomatous Trichiasis Surgery (FLAME) Trial: Study Design. medRxiv [Preprint]. 2024 Jul 7:2024.06.26.24308549. doi: 10.1101/2024.06.26.24308549. PMID 39006430